CLINICAL TRIAL: NCT00139425
Title: Osteoporosis Prevention and Treatment Program: A Disease Management Demonstration Project
Brief Title: Osteoporosis Disease Management Demonstration Project (0000-037)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 0000-037; 037; 2005_048
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

INTERVENTIONS:
Behavioral: Disease Management Assessment

SUMMARY:
The purpose of this study is to assess the impact of disease management interventions on bone mineral density (BMD) screening rates and osteoporosis treatment rates in women age 65 years or older.

ELIGIBILITY:
Inclusion Criteria:

* Members of the Henry Ford Health System

Exclusion Criteria:

* Individuals who are not members of the Henry Ford Health System

Ages: 65 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 10000
Dates: Start 2003-05; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Bone mineral density (BMD) testing rates

SECONDARY OUTCOMES:
Osteoporosis medication treatment rates

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Lafata JE, Kolk D, Peterson EL, McCarthy BD, Weiss TW, Chen YT, Muma BK. Improving osteoporosis screening: results from a randomized cluster trial. J Gen Intern Med. 2007 Mar;22(3):346-51. doi: 10.1007/s11606-006-0060-9. PMID 17356966